CLINICAL TRIAL: NCT03995082
Title: A Randomized Study of Breast Cancer Patient Engagement With Patient Reported Outcome Measure Survey Results
Brief Title: Breast Cancer Patient Engagement With Patient Reported Outcome Measure Survey
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-2562.cc
Record Dates: First submitted 2019-05-22; First posted 2019-06-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients will receive the results from the PROM survey in graphical form each time they complete a survey.
  Interventions: Other: Patient Reported Outcome Measure Survey result feedback
- Normative Control (No Intervention): These patients will complete the PROM surveys, but will not be presented with the results of the survey.

INTERVENTIONS:
Other: Patient Reported Outcome Measure Survey result feedback — Patients will receive a graph of their results from the PROM survey each time they complete a survey
  Arms: Experimental Group

SUMMARY:
The purpose of this research protocol is to measure Patient Reported Outcome Measures (PROMs) in breast cancer patients. PROM results will be provided to patients and providers and the investigators will evaluate the relationship between patient engagement with PROM results and patient and clinicopathologic variables, utilization of supportive and hospital services, and patient satisfaction with patient-provider communication.

DETAILED DESCRIPTION:
PROM Survey The BREAST-Q survey will be utilized to evaluate PROMs at the designated survey time points. The investigators will utilize the mastectomy and breast conserving therapy pre-operative and post-operative modules dependent on the type of surgery each patient chooses. The BREAST-Q survey has questions that pertain to the following domains: 1. Satisfaction with breasts, 2. Psychosocial well-being, 3. Physical well-being, 4. Sexual well-being, 5. Adverse effects of radiation, and 6. Patient experience with the health care team. Scores for each domain are scored with an equivalent Rasch transformed score (range 0-100). These scores can then be tracked over time. In addition to the BREAST-Q modules, the investigators will ask 3 open ended questions. These questions will allow patients to share concerns or outcomes at each time point in an effort to identify currently unmeasured outcomes that are important to patients.

Timing of Surveys For patients having surgery first: At the pre-operative visit, patients will be provided the pre-operative module. The post-operative modules will then be administered via email or in the clinic at the post-operative visit (~2 weeks after surgery), and then at 3 months, 6 months, 9 months, and 12 months after surgery. After one year, patients will be surveyed annually.

For patients receiving neoadjuvant chemotherapy, surveys will be administered every 3 months during the pre-operative period. The post-operative modules will then be administered via email or in the clinic at the post-operative visit (~2 weeks after surgery), and then at 3 months, 6 months, 9 months, and 12 months after surgery. After one year, patients will be surveyed annually.

Patients will be randomized to receive the results of PROM surveys graphed over time (experimental group) or to not receive the results of the PROM surveys (normative control group). Results of the BREAST-Q surveys will be available to providers for all patients.

Statistical Analyses Study data will be collected in a prospective database using the CCTSI RedCap database, with which the breast cancer program has extensive experience. The database will include demographic information, clinicopathologic data, surgical details, neoadjuvant and adjuvant treatments, and the equivalent Rasch transformed scores for each PROM metric at all recorded time points.

Descriptive statistics will be utilized to characterize the patient population and patient engagement with PROMs. Univariate and multivariate analyses will be used to evaluate demographic and clinicopathologic variables and variations in PROMs across the course of treatment. The study endpoints will be evaluated with the following statistical methods:

ELIGIBILITY:
We will target all patients with a new diagnosis of breast cancer who present to the breast multi-disciplinary clinic.

Inclusion:

* Adult (18 years of age or more)
* Female
* Patients with breast cancer
* Patients who can independently complete surveys

Exclusion

* Age <18 years
* Male
* Patients who cannot independently complete surveys

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 925 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
BREAST Q patient satisfaction with breast surgeon domain | 24 months
  Patient satisfaction with patient-provider communication using the BREAST Q satisfaction with breast surgeon domain. The domain is scored from 0 to 100 points with more points representing higher patient satisfaction.

SECONDARY OUTCOMES:
BREAST Q Patient reported outcome measure survey domains including: Satisfaction with breasts, psychosocial well being, physical well being, sexual well being, and effects of radiation domains. | 24 months
  Validated BREAST Q survey domains. All domains are scored 0 to 100 points. Higher points represent a better outcome. The subscales will not be used to create a total score.
Healthcare utilization including the use of social work services, psycho-oncology services, oncology fitness service, nutrition service, and urgent/emergent services including visits to urgent care or the emergency room. | 24 months
  The number of participants using supportive services will be scored as yes or no if the patient used the specific service or did not use the service.
Currently unmeasured patient reported outcomes using open ended questions | 24 months
  The investigators will use open ended questions to identify currently unmeasured patient reported outcomes. Responses will be evaluated as qualitative data using descriptive coding to identify themes. Expected common themes include financial concerns, concerns about caring for family or imposing on family, fertility concerns, etc. The questions will include: "what are your top 3 concerns", "what are you most worried about going forward", "how could the healthcare team better help you", "if you could start your treatment over what would you have done differently."

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Denver, Colorado
  - Cherry Creek Medical Center, Denver, Colorado
  - Lone Tree Medical Center, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No